CLINICAL TRIAL: NCT02467634
Title: A Phase II Proof-of-Concept Study of the Safety and Efficacy of HUCNS-SC Subretinal Transplantation in Subjects With Geographic Atrophy of Age-Related Macular Degeneration
Brief Title: Study of HUCNS-SC Subretinal Transplantation in Subjects With GA of AMD
Acronym: RADIANT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on a business decision unrelated to any safety concerns.
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-AMD-201
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC (Experimental): HuCNS-SC sub-retinal transplantation
  Interventions: Biological: HuCNS-SC sub-retinal transplantation

INTERVENTIONS:
Biological: HuCNS-SC sub-retinal transplantation — HuCNS-SC sub-retinal transplantation in subjects with bilateral GA AMD

SUMMARY:
A fellow eye controlled study of HUCNS-SC sub-retinal transplantation in subjects with bilateral GA AMD. All subjects will be assigned to HUCNS-SC transplantation.

DETAILED DESCRIPTION:
A fellow eye controlled study of HUCNS-SC sub-retinal transplantation in subjects with bilateral geographic atrophy (GA) age-related macular degeneration (AMD). All subjects will be assigned to HUCNS-SC transplantation. All subjects will be followed for efficacy and safety for 12 months. An independent data monitoring committee (IDMC) will review adverse events for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* GA associated with AMD in both eyes. Total area of GA determined by fundus autofluorescence.
* BCVA of 20/320 or better in each eye at screening assessment

Exclusion Criteria:

* Prior or concurrent choroidal neovascularization in either eye by clinical exam and/or fluorescein angiography as determined by the investigator or the reading center.
* Retinal or macular disease of any other cause in either eye.
* Diagnosis of glaucoma in either eye.
* Uncontrolled intraocular pressure in either eye
* Compromised renal function defined as eGFR <60mL/min and urine protein-to-creatinine ration >0.3 is spot urine collection.
* History of or active autoimmune disease.
* Previous organ, tissue or bone marrow transplantation.
* Seropositive for HIV, hepatitis B or C, or CMV IgM

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
GA area based on fundus autofluorescence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, MD, Study Chair — StemCells, Inc.
Locations (12):
- United States (12):
  - Retina Associates Southwest, PC, Tucson, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Research Institute of Texas, Palo Alto, California
  - Rush University Med Ctr., Chicago, Illinois
  - William Beaumont Health System, Royal Oak, Michigan
  - New York Eye and Ear Infirmary, New York, New York
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Research Center, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - University Of Utah / John A. Moran Eye Center, Salt Lake City, Utah